CLINICAL TRIAL: NCT00232596
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Phase 3 Study to Determine the Efficacy and Safety of Retigabine (1200 mg/Day) Used as Adjunctive Therapy in Refractory Epilepsy Patients With Partial-Onset Seizures
Brief Title: Retigabine (Adjunctive Therapy) Efficacy and Safety Study for Partial Onset Refractory Seizures in Epilepsy
Acronym: RESTORE1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VRX-RET-E22-301
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Seizures
Keywords: Partial Seizures; Anticonvulsant; Complex Partial Seizures; Potassium Channels; Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Retigabine (Experimental)
  Interventions: Drug: Retigabine

INTERVENTIONS:
Drug: Retigabine — Oral tablet. The starting daily dose will be 300 mg/day administered orally in three equally divided doses. This dosage will be increased by 150 mg/day (50 mg/dose) at 1-week intervals (titration phase). At the beginning of Week 7, patients will enter a 12 week maintenance phase
  Other Names: D-23129; GKE-841
  Arms: Retigabine
Drug: Placebo — Oral tablet.
  Arms: Placebo

SUMMARY:
This Phase 3 study is being conducted to evaluate the efficacy and safety of retigabine dosed at 1200 mg/day, in three equally divided doses, compared with placebo in patients with epilepsy who are receiving up to three established antiepileptic drugs (AEDs).

DETAILED DESCRIPTION:
This Phase 3 study is being conducted in North America, Argentina, and Brazil to evaluate the efficacy and safety of retigabine dosed at 1200 mg/day, in three equally divided doses, compared with placebo in patients with epilepsy who are receiving up to three established antiepileptic drugs (AEDs). The primary objective is to demonstrate a superior change in total partial seizure frequency for four weeks from baseline to the double-blind period. The proportion of responders (greater than or equal to 50% reduction in total partial seizure frequency for four weeks from baseline to the double-blind period) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory epilepsy with simple or complex partial onset seizures with or without secondary generalization
* 28-day partial seizure frequency rate of four or more partial seizures over the 8-week baseline phase
* Currently treated with up to three established AEDs
* Vagal Nerve Stimulator may be included

Exclusion Criteria:

* Existing medical or psychiatric condition which could affect patient's health or compromise ability to participate in the study
* Clinically significant abnormalities on physical exam, vital signs, ECG, or liver function tests
* Impaired renal function (creatinine clearance less than 50 mL/minute)
* Evidence of progressive central nervous disease, lesion, or encephalopathy
* History of primary generalized seizures
* History of clustering or flurries or status epilepticus within 12 months of study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- United States (32):
  - University of Alabama -- Department of Neurology/Epilepsy Center, Birmingham, Alabama
  - North Alabama Neuroscience Research Associates, Huntsville, Alabama
  - Neurology Clinic, Northport, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Clinical Trials Inc., Little Rock, Arkansas
  - UCSD Thornton Hospital, La Jolla, California
  - University of Southern California, Los Angeles, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - Delta Waves, Colorado Springs, Colorado
  - University of Colorado Health Science Center, Denver, Colorado
  - University of Florida -- Shands Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - McFarland Clinic, Ames, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Epilepsy Group, P.A., Saint Paul, Minnesota
  - The Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Beth Israel Medical Center, New York, New York
  - Asheville Neurology Specialists, Asheville, North Carolina
  - Medical University of Ohio at Toledo, Toledo, Ohio
  - Oregon Neurology PC, Tualatin, Oregon
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Neurological Clinic of Texas, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Virginia Comprehensive Epilepsy Program, Charlottesville, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Argentina (6):
  - Hospital Italiano de Buenos Aires, Capital Federal, CBA
  - Hospital General de Agudos "Dr. J.M. Ramos Mejia", Capital Federal, CBA
  - Hospital General de Agudos "Dr. Teodoro Alvarez", Capital Federal, CBA
  - Fundacion Lennox, Córdoba, CRD
  - Sanatorio del Salvador II, Córdoba, CRD
  - Hospital Privado Centro Medico de Cordoba, Córdoba, CRD
- Brazil (4):
  - Hospital Universitario Prof Edgard Santos -- UFBA, Salvador, Estado de Bahia
  - Hospital das Clinicas de Ribeirao Preto -- Universidade de Sa Neurologia, Ribeirão Preto, São Paulo
  - Hospital Sao Paulo -- Escola Paulista de Medicina -- UNIFESP, São Paulo, São Paulo
  - Hospital das Clinicas da Fac de Medicina de Sao Paulo, São Paulo, São Paulo
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - Glenrose Rehabilitation Center, Edmonton, Alberta
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - CHUM -- Hôpital Notre-Dame, Montreal, Quebec
- Mexico (8):
  - Antiguo Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Instituto Nacional de Neurologia y Neurocirugia, La Fama, Mexico City
  - Centro Medico, Mexico City, Mexico City
  - Hospital de Psiquiatria San Fernando, IMSS, Mexico City, Mexico City
  - CIF BIOTEC, Medica Sur, Tlalpan, Mexico City
  - Hospital y Clinica OCA S.A. de C.V., Monterrey, Nuevo León
  - Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City, San Luis Potosí
  - instituto Nacional de Neurologia y Neurocirugia, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Porter RJ, Burdette DE, Gil-Nagel A, Hall ST, White R, Shaikh S, DeRossett SE. Retigabine as adjunctive therapy in adults with partial-onset seizures: integrated analysis of three pivotal controlled trials. Epilepsy Res. 2012 Aug;101(1-2):103-12. doi: 10.1016/j.eplepsyres.2012.03.010. Epub 2012 Apr 16. PMID 22512894
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: VRX-RET-E22-301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: VRX-RET-E22-301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: VRX-RET-E22-301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: VRX-RET-E22-301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: VRX-RET-E22-301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: VRX-RET-E22-301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: VRX-RET-E22-301 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the Double-blind Phase (Titration plus Maintenance Phases) who elected to continue in the Open-Label Extension Study (OLE-S) entered the Transition Phase, for titration, if on placebo, or to maintain the blind if on retigabine. Participants who did not enter the Titration Phase entered a Taper Phase.
Groups:
- Placebo: Titration Phase: matching placebo tablets of dummy strengths of 50 milligrams (mg), 100 mg, and 300 mg administered orally thrice a day (TID) for 6 weeks. Maintenance Phase: matching placebo tablets of dummy strengths of 50 mg, 100 mg, and 300 mg administered orally TID for 12 weeks.
- Retigabine: Titration Phase: retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID with a starting daily dose of 300 mg/day (in 3 equally divided doses). The dose increased weekly by 150 mg/day (50 mg TID) for the 6 weeks of the Titration Phase to a target daily dose of 1200 mg/day (400 mg TID) by the beginning of Week 7 of treatment. Maintenance Phase: Retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a target daily dose of 1200 mg/day (400 mg TID) for 12 weeks in participants who tolerated this dose. Participants who could not tolerate the 1200 mg/day dose were allowed to reduce the dose to 1050 mg/day (350 mg TID) at the end of the first week and then maintain this dose for the remainder of the 12 weeks.
Period: 6-Week Titration Phase
Arm/Group | Placebo | Retigabine
Started | 152 | 154
Completed | 138 | 125
Not Completed | 14 | 29
Not completed — Adverse Event | 6 | 19
Not completed — Failed to Return | 2 | 1
Not completed — Unsatisfactory Response - Efficacy | 1 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — Participant Request Unrelated to Study | 1 | 0
Not completed — Other | 3 | 3
Not completed — Participant Did Not Receive Study Drug | 0 | 1
Period: 12-Week Maintenance Phase
Arm/Group | Placebo | Retigabine
Started | 138 | 125
Completed | 126 (One participant withdrew after being considered a "completer" and is listed as an early withdraw.) | 97
Not Completed | 12 | 28
Not completed — Adverse Event | 7 | 22
Not completed — Unsatisfactory Response -Efficacy | 1 | 2
Not completed — Protocol Violation | 3 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo - Double-blind (DB) Phase (Titration + Maintenance): Matching placebo tablets of dummy strengths of 50 milligrams (mg), 100 mg, and 300 mg administered orally thrice a day (TID) for 18 weeks (6 weeks of Titration Phase and 12 weeks of Maintenance Phase)
- Retigabine - DB Phase (Titration + Maintenance): Retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a target daily dose of 1200 mg/day (400 mg TID) for 18 weeks (6 weeks of Titration Phase, with dosage increase from 300 mg/day to 1200 mg/day [weekly increase of 150 mg/day], and 12 weeks of Maintenance Phase, with 1200 mg/day or 1050 mg/day [for participants who could not tolerate 1200 mg/day])
- Total: Total of all reporting groups
Arm/Group | Placebo - Double-blind (DB) Phase (Titration + Maintenance) | Retigabine - DB Phase (Titration + Maintenance) | Total
Number analyzed (Participants) | 152 | 153 | 305
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected in the Safety Population, comprised of all participants who received at least one dose of study medication. One participant randomized to the Retigabine group did not receive study medication in the 6-week Titration Phase.
  Years | 36.7 (11.63) | 37.7 (12.55) | 37.2 (12.09)
Gender [Count of Participants; unit: Participants] — Baseline characteristics were collected in the Safety Population, comprised of all participants who received at least one dose of study medication. One participant randomized to the Retigabine group did not receive study medication in the 6-week Titration Phase.
  Participants
    Female | 80 | 85 | 165
    Male | 72 | 68 | 140
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in the Safety Population, comprised of all participants who received at least one dose of study medication. One participant randomized to the Retigabine group did not receive study medication in the 6-week Titration Phase.
  participants
    Caucasian | 78 | 90 | 168
    African - American (Black) | 15 | 15 | 30
    Hispanic | 48 | 39 | 87
    Asian | 1 | 1 | 2
    American Indian | 1 | 0 | 1
    Mestizo | 1 | 0 | 1
    Mixed Race | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the 28-day Total Partial Seizure (PS) Frequency From Baseline (BL) to the End of the Double-blind (DB) Phase (Titration and Maintenance Phases)
Description: 28-day total PS (PSs [also called focal seizures] are seizures limited to a specific area of the brain) frequency in the BL period = (Number [No.] of total PSs reported in the BL period divided by the No. of days of available total PS data in the BL period) x 28 days. 28-day total PS frequency in the DB period = (No. of total PSs reported in the DB period divided by the No. of days of available total PS data in the DB period) x 28 days. Percent change = ([value in the DB period minus value at BL] divided by the BL value) x 100%. Negative values indicate a reduction in seizure frequency.
Time Frame: Baseline (Week -7 through Week 0), Week 1 through Week 18
Population: Intent-to-Treat (ITT) Population for Food and Drug Administration (FDA) review: all randomized participants (par.) who received at least one dose of the study drug. Only par. with baseline and post-baseline measures were analyzed. Two par. in each treatment arm did not have post-baseline measures and were thus not included in this analysis.
Measure: Median (Full Range); unit: percent change in seizure frequency
Groups:
- Placebo - DB Phase (Titration + Maintenance): Matching placebo tablets of dummy strengths of 50 mg, 100 mg, and 300 mg administered orally TID for 18 weeks (6 weeks of Titration Phase and 12 weeks of Maintenance Phase)
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine - DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 150 | 151
percent change in seizure frequency | -17.5 [-90 to 628] | -44.3 [-100 to 302]
Statistical Analysis 1: Comparison: Placebo - DB Phase (Titration + Maintenance) vs Retigabine - DB Phase (Titration + Maintenance); Test type: Superiority or Other; p < 0.001, Non-parametric rank ANCOVA — Non-parametric rank analysis of covariance adjusted for baseline 28-seizure frequency and stratified by baseline seizure frequency category and region

2. Primary Outcome: Number of Participants Who Were Responders and Non-responders in the Maintenance Phase
Description: Responders were participants with at least a 50% reduction in the 28-day total partial seizure frequency in the Maintenance Phase as compared to the Baseline period.
Time Frame: Week 7 through Week 18
Population: Intent-to-Treat (ITT) Population for European Medicines Agency (EMEA) review: all randomized participants who received at least one dose of study drug in the Maintenance Phase and had at least one seizure measurement (whether or not they had a seizure) recorded in the Maintenance Phase
Measure: Number; unit: participants
Groups:
- Placebo - Maintenance Phase: Matching placebo tablets of dummy strengths of 50 mg, 100 mg, and 300 mg administered orally TID for 12 weeks
- Retigabine - Maintenance Phase: Retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a target daily dose of 1200 mg/day (400 mg TID) for 12 weeks of Maintenance Phase, with 1200 mg/day or 1050 mg/day [for participants who could not tolerate 1200 mg/day])
Arm/Group | Placebo - Maintenance Phase | Retigabine - Maintenance Phase
Number analyzed (Participants) | 137 | 119
participants
  Responders | 31 | 66
  Non-responders | 106 | 53
Statistical Analysis 1: Comparison: Placebo - Maintenance Phase vs Retigabine - Maintenance Phase; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Number of Participants Who Were Responders and Non-responders in the DB Phase
Description: Responders were participants with at least a 50% reduction in the 28-day total partial seizure frequency in the DB Phase as compared to the Baseline period. Participants without any post-baseline data were considered non-responders.
Time Frame: Week 1 through Week 18
Population: ITT Population for FDA review
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine - DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 152 | 153
participants
  Responders | 27 | 68
  Non-responders | 125 | 85

4. Secondary Outcome: Percent Change From Baseline (BL) in the 28-day Total Partial Seizure Frequency During the Maintenance Phase
Description: 28-day total partial seizure frequency in the BL period = (No. of total partial seizures reported in the BL period divided by the No. of days of available total partial seizure data in the BL period) x 28 days. 28-day total partial seizure frequency in the Maintenance Phase = (No. of total partial seizures reported in the Maintenance Phase divided by the No. of days of available total partial seizure data in the same phase) x 28 days. Percent change = (value in the Maintenance Phase minus value at BL divided by the BL value) x 100%. Negative values indicate a reduction in seizure frequency.
Time Frame: Baseline (Week -7 through Week 0), Week 7 through Week 18
Population: ITT Population for EMEA review
Measure: Median (Full Range); unit: percent change in seizure frequency
Groups:
- Retigabine - Maintenance Phase: Retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a target daily dose of 1200 mg/day (400 mg TID), for 12 weeks of Maintenance Phase, with 1200 mg/day or 1050 mg/day [for participants who could not tolerate 1200 mg/day])
Arm/Group | Placebo - Maintenance Phase | Retigabine - Maintenance Phase
Number analyzed (Participants) | 137 | 119
percent change in seizure frequency | -18.9 [-100 to 1382] | -54.5 [-100 to 660]

5. Secondary Outcome: Number of Participants With a Reduction in the 28-day Total Partial Seizure Frequency From Baseline to the End of DB Phase (Titration and Maintenance Phases) by Indicated Quartile Reduction Categories
Description: Participants who experienced a reduction from Baseline in the 28-day total partial seizure frequency were categorized as having a reduction of 75-100%, 50-<75%, 25-<50%, or <25%, in addition to having no reduction. This quartile cutting was specified in the study protocol. Participants without any post-baseline data were included in the "No reduction" category.
Time Frame: Baseline (Week -7 through Week 0), Week 1 through Week 18
Population: ITT Population for FDA review
Measure: Number; unit: participants
Groups:
- Retigabine DB Phase (Titration + Maintenance): Retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a target daily dose of 1200 mg/day (400 mg TID) for 18 weeks (6 weeks of Titration Phase, with dosage increase from 300 mg/day to 1200 mg/day [weekly increase of 150 mg/day], and 12 weeks of Maintenance Phase, with 1200 mg/day or 1050 mg/day [for participants who could not tolerate 1200 mg/day])
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 152 | 153
participants
  75% to 100% reduction | 6 | 27
  50% to <75% reduction | 21 | 41
  25% to <50% reduction | 37 | 20
  >0 to <25% reduction | 33 | 26
  No reduction | 55 | 39

6. Secondary Outcome: Number of Participants With a Reduction in the 28-day Total Partial Seizure Frequency From Baseline to the End of the DB Phase (Titration and Maintenance Phases) by Indicated Decile Reduction and Increase Categories
Description: Participants who experienced a reduction from Baseline in the 28-day total partial seizure frequency were categorized in decile cutting, i.e., reduction categories of 90-100%, 80-<90%, 70-<80%, 60-<70%, 50-<60%, 40-<50%, 30-<40%, 20-<30%, 10-<20%, >0-<10%, and increase categories of 0-10%, >10-20%, >20-30%, >30% (FDA endpoint). Participants without any post-baseline data were included in the 0-10% increase category.
Time Frame: Baseline (Week -7 through Week 0), Week 1 through Week 18
Population: ITT Population for FDA review
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 152 | 153
participants
  Reduction: 90% to 100% | 0 | 12
  Reduction: 80% to <90% | 5 | 11
  Reduction: 70% to <80% | 4 | 10
  Reduction: 60% to <70% | 7 | 20
  Reduction: 50% to <60% | 11 | 15
  Reduction: 40% to <50% | 11 | 10
  Reduction: 30% to <40% | 13 | 6
  Reduction: 20% to <30% | 19 | 12
  Reduction: 10% to <20% | 13 | 10
  Reduction: >0% to <10% | 14 | 8
  Increase: 0% to 10% | 14 | 10
  Increase: >10% to 20% | 12 | 5
  Increase: >20% to 30% | 4 | 4
  Increase: >30% | 25 | 20

7. Secondary Outcome: Number of Participants With the Indicated Reduction From Baseline in the 28-day Total Partial Seizure Frequency During the Maintenance Phase
Description: Participants who experienced a reduction from Baseline in the 28-day total partial seizure frequency were categorized as having a >75%, a 50-75%, or a <50% reduction, in addition to having no reduction (EMEA endpoint).
Time Frame: Baseline (Week -7 through Week 0), Week 7 through Week 18
Population: ITT Population for EMEA review
Measure: Number; unit: participants
Arm/Group | Placebo - Maintenance Phase | Retigabine - Maintenance Phase
Number analyzed (Participants) | 137 | 119
participants
  >75% reduction | 13 | 37
  50% to 75% reduction | 18 | 29
  >0 to <50% reduction | 65 | 33
  No reduction | 41 | 20

8. Secondary Outcome: Number of Participants Who Experienced the Indicated Level of Exacerbation and Reduction in the 28-day Total Partial Seizure Frequency From Baseline During the Maintenance Phase
Description: Participants who experienced an exacerbation from Baseline in the 28-day total partial seizure frequency were categorized as having a 0-25% or a >25% increase (EMEA endpoint). The number of participants experiencing a >0% reduction from Baseline in the 28-day total partial seizure frequency are also presented.
Time Frame: Baseline (Week -7 through Week 0), Week 7 through Week 18
Population: ITT Population for EMEA review.
Measure: Number; unit: participants
Arm/Group | Placebo - Maintenance Phase | Retigabine - Maintenance Phase
Number analyzed (Participants) | 137 | 119
participants
  0% to 25% increase | 20 | 4
  >=25% increase | 21 | 16
  >0% reduction | 96 | 99

9. Secondary Outcome: Number of Participants Reporting New Seizure Types in the Indicated Categories During the DB Phase (Titration and Maintenance Phases) That Were Not Reported at Baseline
Description: New seizure types included those seizures which were not reported by any participant at Baseline.
Time Frame: Baseline (Week -7 through Week 0), Week 1 through Week 18
Population: ITT Population for FDA review
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 152 | 153
participants
  No new seizure type | 33 | 42
  Partial seizures without motor signs | 12 | 17
  Partial evolving to secondarily generalized | 7 | 12
  Complex partial seizures | 5 | 11
  Partial seizures with motor signs | 11 | 7
  Flurries | 3 | 1
  Tonic-clonic seizures | 0 | 1
  Atonic seizures | 1 | 0

10. Secondary Outcome: Number of Participants Who Were Seizure-free During the DB Phase (Titration and Maintenance Phases)
Description: Participants were considered to be seizure-free if they had not reported any seizures during the DB treatment period (Weeks 1-18). For a participant to be seizure free during the DB Phase, the participant had to be seizure free both Week 7 to Week 18 and Week 1 to Week 6. A participant could be seizure free Week 7 to Week 18 (during the Maintenance Phase), but not seizure free Week 1 to Week 6. Hence, there are fewer participants being reported as seizure free from Week 1 to Week 18 than from Week 7 to Week 18.
Time Frame: Week 1 through Week 18
Population: ITT Population for FDA review. Only participants who had post-baseline seizure data were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 150 | 151
participants
  Seizure free | 0 | 3
  Not seizure free | 150 | 148

11. Secondary Outcome: Number of Participants Who Were Seizure-free During the Maintenance Phase
Description: Participants were considered to be seizure-free if they had not reported any seizures during the Maintenance Phase.
Time Frame: Week 7 through Week 18
Population: ITT Population for EMEA review
Measure: Number; unit: participants
Arm/Group | Placebo - Maintenance Phase | Retigabine - Maintenance Phase
Number analyzed (Participants) | 137 | 119
participants
  Seizure free | 2 | 9
  Not seizure free | 135 | 110

12. Secondary Outcome: Percentage of Seizure-free Days During the DB Phase (Titration and Maintenance Phases)
Description: A seizure-free day was a day without any seizures. For a participant to be seizure free during the DB Phase, the participant had to be seizure free both Week 7 to Week 18 and Week 1 to Week 6. A participant could be seizure free Week 7 to Week 18 (during the Maintenance Phase), but not seizure free Week 1 to Week 6. Hence, there are fewer participants being reported as seizure free from Week 1 to Week 18 than from Week 7 to Week 18. The percentage of seizure-free days was calculated as the total number of days without seizures in the DB period divided by the number of days in DB period x 100%.
Time Frame: Week 1 through Week 18
Population: ITT Population for FDA review. Only participants who had post-baseline seizure data were included in the analysis.
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 150 | 151
percentage of days | 77.3 [0 to 98] | 84.1 [0 to 100]

13. Secondary Outcome: Percentage of Seizure-free Days During the Maintenance Phase
Description: A seizure-free day was a day without any seizures. The percentage of seizure-free days was calculated as the total number of days without seizures in the DB period divided by the number of days in the DB period x 100%.
Time Frame: Week 7 through Week 18
Population: ITT Population for EMEA review
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Placebo - Maintenance Phase | Retigabine - Maintenance Phase
Number analyzed (Participants) | 137 | 119
percentage of days | 78.2 [0 to 100] | 86.9 [0 to 100]

14. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at the End of the Maintenance Phase
Description: Clinical Global Impression of Improvement (CGI-I) is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the treatment. Scores on the scale are rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Week 18/end of treatment phase
Population: ITT Population for EMEA review. Only participants who had CGI-I scores were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo - Maintenance Phase | Retigabine - Maintenance Phase
Number analyzed (Participants) | 137 | 117
scores on a scale | 3.2 (1.11) | 2.7 (1.30)

15. Secondary Outcome: Patient Global Impression (PGI) Score at the End of the Maintenance Phase
Description: PGI is a participant-rated scale of improvement that was administered at the end of the Maintenance Phase in order to assess the participant's impression of his or her own improvement. PGI assessments were scored using a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: Week 18/end of treatment phase
Population: ITT Population for EMEA review. Only participants who had a PGI score were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo - Maintenance Phase | Retigabine - Maintenance Phase
Number analyzed (Participants) | 120 | 100
scores on a scale | 2.9 (1.16) | 2.9 (1.23)

16. Secondary Outcome: Quality of Life (QOL) Assessed by QOL in Epilepsy-Problems Questionnaire (QOLIE-31-P) at Baseline (Week 0) and Weeks 6, 10, and 18
Description: The QOLIE-31-P is a 31-item questionnaire evaluating a participant's QOL perception in 7 domains: seizure worry, emotional well being, energy/fatigue, cognitive functioning, medication effects, social functioning, overall QOL. Precoded numeric values for some domains are such that a higher number reflects a more favorable health state; others are such that a higher number reflects a less favorable state. Precoded values are first converted to 0-100 point scores; higher converted scores always reflect better QOL. The overall score is derived by weighting and then summing the 7 domain scores.
Time Frame: End of Baseline (Week 0), Weeks 6, 10, and 18
Population: Safety Population: all randomized participants who received at least 1 dose of retigabine or placebo. Participants who were cognitively impaired and could not complete the QOLIE-31-P assessment were not analyzed. The number of participants analyzed differs by week because not all participants completed the questionnaire at the indicated weeks.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 139 | 137
scores on a scale
  Baseline (Week -7 through Week 0), n=139, 137 | 52.6 (15.55) | 55.6 (17.95)
  Week 6 (Titration Phase), n=127, 108 | 55.2 (16.71) | 55.7 (19.18)
  Week 10 (Maintenance Phase), n=121, 102 | 57.9 (15.57) | 56.2 (18.04)
  Week 18 (Maintenance Phase), n=116, 85 | 57.3 (15.56) | 53.8 (17.79)

17. Secondary Outcome: Number of Participants Whose Clinical Laboratory Values Were Deemed an Adverse Event by the Investigator (>=2% in Any Treatment Arm)
Description: Clinically important changes in laboratory values were to be reported as an adverse event if they met one of the following criteria: (1) intervention required; (2) change in dose of study drug required; (3) other treatment/therapy required; (4) association with other diagnoses.
Time Frame: Week 1 through Week 24
Population: Safety Population
Measure: Number; unit: participants
Groups:
- Placebo - DB Phase (Titration and Maintenance): Matching placebo tablets of dummy strengths of 50 mg, 100 mg, and 300 mg administered orally TID for 18 weeks (6 weeks of Titration Phase and 12 weeks of Maintenance Phase)
- Placebo (DB Phase) and Retigabine (Transition Phase): Participants on placebo during the DB phase were administered retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a total daily dose of 1200 mg/day (400 mg TID) for 6 weeks
- Retigabine - DB Phase (Titration and Maintenance): Retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a target daily dose of 1200 mg/day (400 mg TID) for 18 weeks (6 weeks of the Titration Phase, with dosage increase from 300 mg/day to 1200 mg/day [weekly increase of 150 mg/day], and 12 weeks of the Maintenance Phase, with 1200 mg/day or 1050 mg/day [for participants who could not tolerate 1200 mg/day])
- Retigabine (DB Phase) and Retigabine (Transition Phase): Participants on retigabine during the DB phase were administered retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a total daily dose of 1200 mg/day (400 mg TID) for 6 weeks
Arm/Group | Placebo - DB Phase (Titration and Maintenance) | Placebo (DB Phase) and Retigabine (Transition Phase) | Retigabine - DB Phase (Titration and Maintenance) | Retigabine (DB Phase) and Retigabine (Transition Phase)
Number analyzed (Participants) | 152 | 123 | 153 | 92
participants
  Urine analysis abnormal | 3 | 3 | 4 | 2
  Bacteria urine | 1 | 0 | 1 | 2
  Hematology test abnormal | 0 | 0 | 1 | 2
  Urinary sediment present | 1 | 0 | 0 | 2

18. Secondary Outcome: Number of Participants Who Reported the Indicated Renal and Urinary Disorder Adverse Events at a Frequency Threshold of 2% (in Any Treatment Arm)
Description: A summary of the adverse events classified as renal or urinary disorders and in which at least 2% (rounded to an integer) of participants in any treatment arm reported during the study is presented.
Time Frame: Week 1 through Week 24
Population: Safety Population
Measure: Number; unit: participants
Groups:
- Retigabine - DB Phase (Titration and Maintenance): Retigabine tablets of strengths 50 mg, 100 mg, and 300 mg administered orally TID for a target daily dose of 1200 mg/day (400 mg TID) for 18 weeks (6 weeks of Titration Phase, with dosage increase from 300 mg/day to 1200 mg/day [weekly increase of 150 mg/day], and 12 weeks of Maintenance Phase, with 1200 mg/day or 1050 mg/day [for participants who could not tolerate 1200 mg/day])
Arm/Group | Placebo - DB Phase (Titration and Maintenance) | Placebo (DB Phase) and Retigabine (Transition Phase) | Retigabine - DB Phase (Titration and Maintenance) | Retigabine (DB Phase) and Retigabine (Transition Phase)
Number analyzed (Participants) | 152 | 123 | 153 | 92
participants
  Urinary hesitation | 1 | 2 | 9 | 0
  Dysuria | 2 | 2 | 8 | 1
  Chromaturia | 0 | 0 | 7 | 0
  Polyuria | 1 | 0 | 4 | 0
  Nephrolithiasis | 0 | 0 | 4 | 0
  Hematuria | 1 | 2 | 2 | 0
  Urinary retention | 2 | 2 | 1 | 0

19. Secondary Outcome: Change From Baseline in Post-void Residual Urine Volume at Weeks 10 and 18 of the DB Treatment Phase
Description: Post-void residual (PVR) urine refers to the amount of urine remaining in the bladder after normal urination. To investigate the possible effects of retigabine on bladder function, all participants underwent post-void residual bladder ultrasound at Baseline and during the Maintenance Phase. The PVR bladder ultrasound was performed by a urologist, a qualified ultrasound technician, or a qualified study nurse who was certified to do PVR bladder ultrasound. Change from Baseline in PVR residual volume was calculated as the values at Week 10 and Week 18 minus the value at Baseline.
Time Frame: Baseline (Week -7 through Week 0), Weeks 10 and 18
Population: Safety Population. Only participants who remained in the study at the indicated week and who also had a PVR assessment were analyzed.
Measure: Median (Full Range); unit: milliliters
Arm/Group | Placebo - DB Phase (Titration and Maintenance) | Retigabine - DB Phase (Titration and Maintenance)
Number analyzed (Participants) | 111 | 100
milliliters
  Week 10, n=111, 100 | -1.0 [-211 to 190] | 0.0 [-163 to 413]
  Week 18, n=95, 76 | -3.0 [-258 to 110] | 0.0 [-184 to 257]

20. Secondary Outcome: Number of Participants With a >=7% Increase in Body Weight During Weeks 2, 4, and 6 of theTitration Phase and Weeks 7, 8, 10, 14, and 18 of the Maintenance Phase
Description: The number of participants with recorded weight gain of >=7% over their baseline weight was measured.
Time Frame: Weeks 2, 4, 6 of Titration Phase and Weeks 7, 8, 10, 14, and 18 of Maintenance Phase
Population: Safety Population. Only participants who remained in the study at the indicated week and who also had a body weight assessment were analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo - DB Phase (Titration + Maintenance) | Retigabine DB Phase (Titration + Maintenance)
Number analyzed (Participants) | 149 | 150
participants
  Titration Phase, Week 2, n=149, 150 | 0 | 5
  Titration Phase, Week 4, n=145, 144 | 0 | 5
  Titration Phase, Week 6, n=146, 129 | 1 | 6
  Maintenance Phase, Week 7, n=130, 121 | 2 | 9
  Maintenance Phase, Week 8, n=135, 128 | 1 | 10
  Maintenance Phase, Week 10, n=136, 119 | 3 | 15
  Maintenance Phase, Week 14, n=137, 109 | 3 | 18
  Maintenance Phase, Week 18, n=127, 92 | 4 | 17

ADVERSE EVENTS:
Groups:
- Placebo - Double-blind (DB) Phase (Titration and Maintenance): Matching placebo tablets of dummy strengths of 50 mg, 100 mg, and 300 mg administered orally TID for 18 weeks (6 weeks of Titration Phase and 12 weeks of Maintenance Phase)
Arm/Group | Placebo - Double-blind (DB) Phase (Titration and Maintenance) | Placebo (DB Phase) and Retigabine (Transition Phase) | Retigabine - DB Phase (Titration and Maintenance) | Retigabine (DB Phase) and Retigabine (Transition Phase)
Serious Adverse Events (participants affected / at risk) | 8/152 | 6/123 | 19/153 | 5/92
Other Adverse Events (participants affected / at risk) | 91/152 | 64/123 | 121/153 | 35/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Double-blind (DB) Phase (Titration and Maintenance) (N=152) | Placebo (DB Phase) and Retigabine (Transition Phase) (N=123) | Retigabine - DB Phase (Titration and Maintenance) (N=153) | Retigabine (DB Phase) and Retigabine (Transition Phase) (N=92)
Encephalopathy (Nervous system disorders) | 0 | 0 | 2 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 3 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Device malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Venous Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - Double-blind (DB) Phase (Titration and Maintenance) (N=152) | Placebo (DB Phase) and Retigabine (Transition Phase) (N=123) | Retigabine - DB Phase (Titration and Maintenance) (N=153) | Retigabine (DB Phase) and Retigabine (Transition Phase) (N=92)
Dizziness (Nervous system disorders) | 21 | 19 | 62 | 9
Somnolence (Nervous system disorders) | 27 | 16 | 48 | 5
Fatigue (General disorders) | 12 | 11 | 24 | 1
Confusional state (Psychiatric disorders) | 3 | 4 | 20 | 0
Headache (Nervous system disorders) | 28 | 9 | 19 | 5
Dysarthria (Nervous system disorders) | 3 | 7 | 19 | 0
Urinary tract infection (Infections and infestations) | 13 | 8 | 18 | 4
Ataxia (Nervous system disorders) | 6 | 5 | 17 | 1
Vision blurred (Eye disorders) | 4 | 4 | 18 | 1
Tremor (Nervous system disorders) | 6 | 1 | 17 | 1
Nausea (Gastrointestinal disorders) | 10 | 3 | 16 | 1
Speech disorder (Nervous system disorders) | 0 | 3 | 13 | 2
Influenza (Infections and infestations) | 8 | 3 | 12 | 4
Memory impairment (Nervous system disorders) | 7 | 2 | 12 | 2
Diplopia (Eye disorders) | 4 | 4 | 10 | 0
Gait disturbance (General disorders) | 3 | 4 | 10 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 6 | 9 | 0
Constipation (Gastrointestinal disorders) | 3 | 4 | 9 | 2
Balance disorder (Nervous system disorders) | 1 | 2 | 9 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 2 | 9 | 0
Vomiting (Gastrointestinal disorders) | 8 | 1 | 7 | 0
Anxiety (Psychiatric disorders) | 4 | 6 | 8 | 1
Dysuria (Renal and urinary disorders) | 2 | 2 | 8 | 1
Disorientation (Psychiatric disorders) | 1 | 1 | 8 | 1
Disturbance in attention (Nervous system disorders) | 1 | 4 | 8 | 1
Convulsion (Nervous system disorders) | 9 | 3 | 6 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 2 | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 8 | 3 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.